CLINICAL TRIAL: NCT05300269
Title: SHR-1701 in Combination With Radiotherapy and Chemotherapy as Perioperative Treatment for Resectable Locally Advanced Rectal Cancer, an Open Label, Single-arm, Multicenter Phase II Trial
Brief Title: SHR-1701 in Combination With Chemotherapy and Radiotherapy in Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-II-213
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-03

CONDITIONS: Locally Advanced Rectal Cancer

STUDY DESIGN:
Intervention Model Description: A multicenter, open, single-arm, two-stage phase II clinical study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perioperative treatment (Experimental): Eligible subjects will receive standard chemoradiotherapy with SHR-1701 followed by XELOX combined with SHR-1701 and surgery. Adjuvant XELOX combined with SHR-1701 will be given after surgery.
  Interventions: Drug: SHR-1701；Capecitabine；Oxaliplatin

INTERVENTIONS:
Drug: SHR-1701；Capecitabine；Oxaliplatin — Radiation: Radiation therapy 50.4Gy in 28 fractions to the pelvis on Days 1-5 every week. Drug: Capecitabine Capecitabine 825mg/m^2 orally twice daily (bid) 5 days/week during radiotherapy.
  Drug:SHR-1701 Drug: Capecitabine (XELOX) Capecitabine 1000mg/m^2 orally twice daily (bid) day1-day14, q3w. Drug: Oxaliplatin Oxaliplatin 130mg/m^2, day1, iv, q3w

SUMMARY:
This study will evaluate the efficacy and safety of SHR-1701 combined with radiotherapy and chemotherapy as perioperative treatment for locally advanced rectal cancer. Eligible patients will receive standard chemoradiation with SHR-1701 followed by XELOX combined with SHR-1701. In all subjects, restaging pelvic MRI with chest and abdominal CT will be performed after completion of neoadjuvant treatment to determine resectability and to rule out any evidence of metastases. Subjects who have resectable disease will undergo surgery. Adjuvant XELOX combined with SHR-1701 will be given after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Locally advanced rectal adenocarcinoma and was evaluated as resectable ;
3. The inferior margin of the tumor ≤ 10 cm from the anal verge ;
4. No prior anti-cancer treatment for rectal cancer;
5. Estern Cooperative Oncology Group (ECOG) Performance status (PS) of 0 or 1;
6. Adequate hematologic and end-organ function;
7. Contraception was initiated from the signing of the informed consent until at least 6 months after the last dosing of the study drug

Exclusion Criteria:

1. Unresectable disease determined by investigators
2. Recurrent rectal cancer
3. Evidence of metastatic disease or lateral lymph node metastases
4. Presence of synchronous colorectal cancer
5. Presence of obstruction or imminent obstruction
6. Not eligible for long-course radiotherapy
7. Severe cardiovascular and cerebrovascular diseases;Have clinical heart symptoms or diseases that are not well controlled
8. Prior malignancy within the prior 5 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical/breast cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | At week 16, DAY1
Percentage of participants with Pathological complete response ( pCR ) | At week 16, DAY1

SECONDARY OUTCOMES:
Tumor regression grade ( TRG ) | At week 16, DAY1
Percentage of participants with R0 Resection ( R0 ) | At week 16, DAY1
Percentage of participants with Clinical complete response ( cCR ) rate. | At week 16, DAY1
Event-free survival ( EFS ) | Year 1, Year 2, Year 3
Overall survival ( OS ) | Year 1, Year 2, Year 3
Disease-free survival ( DFS ) | Year 1, Year 2, Year 3

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tang W, Lv Y, Xie H, Wei Y, Wang J, Yu M, Jiang Y, Mao R, Huang C, Rao S, Ding K, Chang W, He G, Xu J. Efficacy and safety of SHR-1701 combined with chemoradiotherapy as neoadjuvant treatment for locally advanced rectal cancer. Cancer Lett. 2026 Jan 1;636:218006. doi: 10.1016/j.canlet.2025.218006. Epub 2025 Aug 26. PMID 40876501